CLINICAL TRIAL: NCT03055364
Title: Observational Study Evaluating Neurocognitive Function in Patients With Primary CNS Malignancy Receiving Radiation Treatment to the Brain
Brief Title: Cognitive Function After Treatment of Primary CNS Malignancy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nadia N. Laack, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 16-005982; NCI-2024-00947 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2017-02-13; First posted 2017-02-16 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: CNS Malignancy
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators propose to evaluate cognitive function and determine the feasibility of neurocognitive assessment using a select CogState test battery in patients with primary intracranial malignancies receiving photon- or proton-based cranial irradiation with curative intent. The investigators will use the CogState software to quantify changes in verbal learning, memory, and executive function over the initial months and years following radiation treatment. Cognitive changes and temporal patterns of function will be compared to baseline performance for each patient. Data regarding cognitive function, fatigue, quality of life, and standard patient reported outcomes will be collected to characterize the daily impact of treatment. In addition, observed outcomes will be correlated with dosimetry values, radiation dose volumes, and anatomic dose distribution.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4 years with primary CNS malignancy
* Able to use computer for assessment battery
* Receiving photon- or proton-based radiation for primary intracranial malignancy
* Demonstrates the capacity to sign informed consent

Exclusion Criteria:

* Patients with WHO Grade IV tumors

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary CNS malignancy
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
characterize the rate and magnitude of change in cognitive performance within 12 months of completion of therapy in patients with intracranial malignancies receiving photon- or proton-based cranial irradiation with curative intent | baseline, completion of treatment, 3 months, 6 months, 1 year and 2 years after radiotherapy
  Using the CogState software

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N. Laack, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials